CLINICAL TRIAL: NCT05317052
Title: From Non-Pharmacologıcal Methods Applied to Primipars in Travay; The Effect of Massage And Music Therapy on Birth Pain, Posttravmatic Comfort and Posttraumatic Development: A Randomized Controlled Study
Brief Title: The Effect of Massage and Musıc Therapy on Birth Pain, Posttravmatic Comfort and Posttraumatic Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Emine Akca, Clinical Researcher of the Amasya University Midwifery Department, Amasya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Amasya U
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Labor Pain; Posttraumatic Growth
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage (Experimental): Massage therapy
  Interventions: Behavioral: Massage group
- Music (Experimental): Music therapy
  Interventions: Behavioral: Massage group
- Control (No Intervention): Control

INTERVENTIONS:
Behavioral: Massage group — Massage and music therapy
  Other Names: Music group
  Arms: Massage; Music

SUMMARY:
Birth pain is the most severe painful experience faced by primiparous people. Massage and music therapy reduce tension in the muscles and reduce the feeling of pain. Massage and music therapy will be applied to pregnant women. No intervention will be made to a group of pregnant women. Numerical Pain Assessment, Post Traumatic Development Scale and Birth Comfort Scale will be used in the research.

DETAILED DESCRIPTION:
Birth pain is one of the most severe and difficult to control pains known. Non-pharmacological methods used to cope with labor pain are cheap and reliable. Massage and music therapy in the first stage of labor are non-pharmacological methods used to reduce labor pain. The purpose of this research; non-pharmacological methods applied to primiparous in labor; The aim of this study is to examine the effects of massage and music therapy on labor pain, postpartum comfort and posttraumatic development. A total of 114 primiparous pregnant women who had a normal delivery expectation and were in the active phase of labor (4-5 cm dilatation) were planned to be included in the study. Massage and music therapy will be applied to pregnant women. No intervention will be made to a group of pregnant women. Numerical Pain Assessment, Post Traumatic Development Scale and Birth Comfort Scale will be used in the research.

ELIGIBILITY:
Inclusion Criteria:

* Expectation of normal vaginal delivery
* Having a term pregnancy
* Being primiparous - Being in the active phase of labor (Cervical dilatation 4 cm)
* Single pregnancy
* Being in vertex presentation
* Uncomplicated prenatal process
* Volunteering to participate in the study
* Being pregnant without back pain

Exclusion Criteria:

* Pregnant women whose birth resulted in cesarean section due to failure of labor to progress during labor
* Pregnant women who did not undergo induction
* Pregnant women who underwent pharmacological intervention for labor pain

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Primiparous pregnant women
Enrollment: 105 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Score | In the labour (active and transition phase)
  The score ranges from 1 to 10 peints, with increasing score reflecting more discomfort

SECONDARY OUTCOMES:
Postpartum Comfort Scale | At the enf of the delivery (In the 24 th hours)
  It is possible to score between 34 and 170 on the scale. An increase in the scores obtained from the scale represents a high level of comfort.
Posttraumatic Growth Inventory | At the enf of the delivery (In the 24 th hours)
  A minimum of 0 and a maximum of 105 points can be obtained from the scale. As the score obtained from the scale increases, it is thought that the level of post-traumatic development is higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No